CLINICAL TRIAL: NCT04663633
Title: The Effect of Eight-week Specific Core Training on Core Stability, Balances and Jumps in Young Rhythmic Gymnasts
Acronym: CST-RG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ramon Llull (Other)
Collaborators: Mònica Solana-Tramunt (Unknown); Jose Morales (Unknown)
Responsible Party: Principal Investigator, Cristina Cabrejas Mata, University professor, University Ramon Llull
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CST-RG
Record Dates: First submitted 2020-11-12; First posted 2020-12-11 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: ATHLETIC PERFORMANCE
Keywords: Core Stability; Core Stability Training; Rhythmic Gymnastics; Plyometric Training; Balance; Rhythmic Gymnastics Jumps

STUDY DESIGN:
Intervention Model Description: Pre-test, intervention and post-test. The Experimental Group performs an eight-week Core Stability Training 3 days a week and the Control Group performs the traditional Rhythmic Gymnastics Training during that period of time.
Who Masked: Outcomes Assessor
Masking Description: The assessment of the test is conducted by masked assessors (judges and physiotherapists)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core stability training (Experimental): The EG performed an 8-week core stability training, consisting in 30 min of core stability and plyometric exercises 3 days per week, 24 sessions in total.
  The CST sessions were conducted in a gym suitable for RG practise and the safety of the participants will be maintained. The equipment necessary for the training was provided to the participants.
  The coaches are RG professionals with national coach level in RG and volunteered to lead the specific CST designed by a RG national coach and an expert core stability physiotherapist.
  Before each session EG and CG performed a 15 min warm up. The load of the session was calculated by the RPE (rate of perceived exertion). And was modulated in order to maintain 7-8 intensity.
  Interventions: Other: Core stability training
- Traditional RG training (No Intervention): The CG performed the traditional training while the EG carried out the CST. The training load was calculated to be 7-8 RPE in order that both groups (EG and CG) undergo an equivalent intensity and training load.

INTERVENTIONS:
Other: Core stability training — Functional Rhythmic Core Stability exercises performed by the experimental group. 30 minutes insert included in the Gymnasts regular training.
  Arms: Core stability training

SUMMARY:
The aim of the study is to evaluate the effect of an eight-week specific Core Stability Training (CST) on young rhythmic gymnasts. The literature suggests CST may help improve sport performance, however, more studies implementing functional CST and accurate methodology are needed to validate this statement. Little is known about Core Stability (CS) and Rhythmic Gymnastics (RG). The study intends to find out whether CST contributes to the Rhythmic gymnasts core stability, balances and jumps execution enhancement, very important RG performance determinants. It is hypothesized the rhythmic gymnasts will increase their CS, balances and jumps performance once the specific CST is conducted.

DETAILED DESCRIPTION:
Gymnasts were recruited from the Gymnastics Club "Gimnàstica Muntanyenc". All participants were rhythmic gymnasts who had at least two-year experience competing in RG at regional federated and school competition level and trained three times per week. Individuals who didn't meet these criteria or were injured at the moment were excluded. The participants were invited to take part in the study voluntarily, and along with their parents were informed verbally and in writing as to the characteristics of the program. Parents or legal guardians signed informed consent forms, and a document that explained the objectives and planned activities of the provided program. The study was approved by the FPCEE Blanquerna Research Ethics Committee. All protocols applied in this research (including the management of the personal data of the participants) complied with the requirements specified in the Declaration of Helsinki of 1975 and its subsequent revisions.

The specific CST program is aimed for Rhythmic gymnasts between 8 and 15 years of age who train in the competitive group and their goal is to improve their RG level. All the study participants were asked to sign an informed consent document that was drafted in keeping with all applicable research ethics protocols, including a guarantee of the confidentiality of personal data and an assurance that participants can choose to abandon the study at any time.

Control group (CG), experimental group (EG) and pre-test, post-test methodology was selected. EG performed the specific CST while CG carried out the traditional RG training.

The CST intervention had been carried out over the course of one academic year (2018-19). The first 3 months allowed investigators to recruit the participants and design the CST adapted to the Rhythmic gymnasts and pursuing the highest specificity for the CS exercises. This design took into account prior experiences of a CS physiotherapist expert and a RG national coach. The load of the sessions was controlled according to a Rate of Perceived Exertion (RPE) scale, a valid method of quantifying exercise training during a wide variety of types of exercise. A training protocol trial will be applied where the subjects will be asked to point out which is their perceived exercise intensity, thirty minutes after the training ends. The repetitions will be adjusted to the 7-8 RPE scale values (very hard) allowing the correct execution of the exercises to the participants and yet permitting adaptations produced by the training. The conclusions drawn from this initial experience formed the scientific basis for the definitive version of the CST.

During the fourth month a pre-test was carried out including an anthropometric study of the gymnasts, three CS tests, seven balance tests and six jump tests. The participants warmed up before each test except for the anthropometric study and the order of the subjects and the order of the applied tests were randomly determined using a true random number generator to avoid order effects. A group blinded specialized physiotherapist conducted the anthropometric study and the CS tests, and a group blinded RG expert led the rest of the tests.

CS tests: Two pressure biofeedback unit (PBU) tests were applied to evaluate the lumbopelvic motor control (LPMC) and the pelvic tilt tests were conducted to evaluate CS endurance.

Balance tests: One leg stand test (OLST) was performed on a force platform to evaluate the gymnasts' balance. Right and left and open and closed eyes conditions were used to perform the four Romberg variants balance tests. Three specific Rhythmic balances were chosen to execute over the force platform and were also evaluated by three RG judge experts.

Jump Tests: Counter movement jump (CMJ) and single leg countermovement jump (SLCMJ) were performed on a force platform to assess the gymnasts' jump. Three specific RG jumps outside the force platform were evaluated by three RG judge experts.

Anthropometric study: A complete anthropometric study was carried out by a professional physiotherapist and will allow the investigators to verify the results are not affected by group initial differences.

From February to April the eight-week CST sessions were offered in the gymnasts' regular training space suitable for the intervention exercises and guaranteeing the safety of the participants. The investigators provided all the extra equipment required for the study. The EG participants performed the CST 3 times per week at the same time of their scheduled training. The duration of the specific training was approximately 30 minutes for 8 weeks with a total of 24 sessions. EG gymnasts were observed while performing the exercises to ensure the training was performed correctly.

Thirty minutes after every CST session all gymnasts (EG and CG) were asked to pick the score of the RPE scale that best described their sensation. This score, multiplied by the minutes of the session (RPE session), helped us modulate the training periodization plan. The average RPE session values were calculated to ensure no load training differences existed among groups.

This CST program involves exercises that challenge the balance, postural control and explosive strength of the gymnasts, executed with specific RG elements and postures.

The specific CST training contains three blocks; a circuit, plyometric exercises and CS exercises. Three different balances and leaps very common in RG (novice to intermediate competitive level) were selected to convert the core and the explosive strength exercises into a very specific and functional training. The balances selected were the passé balance, the side balance with help and the arabesque, the three leaps were the scissors, the stag from assemble and the split leap. The mentioned RG elements were selected due to their lower limb position planes variety and different techniques since it is advised that a range of exercises should be performed to challenge the core musculature in all three planes and ranges of movement to develop total CS. Moreover, all exercises were executed equitably for the right and left side. Unstable superficies as the Bossu, unstable discs and soft balls were included to perform core and balance exercises. The gymnasts performed 3 exercises of the circuit on an unstable surface. It is reported, when standing on an unstable support, the stabilizing muscles make anticipatory adjustments subsequently minimizing postural destabilization. The protocol training and the exercises were conducted by Club Muntanyenc professional RG coaches.

A post-test was performed after the eight-week specific CST following the same procedure as the pre-test.

The Statistical Analysis will be performed using an Excel spreadsheet and then exported to the computer program SPSS statistics 22.0, to then perform the various statistical tests. Initially, a normality test will be performed to check the distribution of the data and to decide whether parametric or non-parametric tests are applied. The G-POWER program will be used to calculate the statistical power of the sample with a value of p <0.05 and an estimated effect size of 0.5.

ELIGIBILITY:
Inclusion Criteria:

* Competition Gymnasts from Club Muntanyenc Sant Cugat training minimum 3 times per week

Exclusion Criteria:

* Injured Gymnasts

Ages: 8 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Core stability results on Lumbo-pelvic motor control (LPMC) | Up to 12 weeks
  Change from pre-test to post-test in LPMC results.
  Active Straight Leg Rise (ASLR) test and Bent Knee Fall Out (BKFO) test are the Pressure Biofeedback Unit (PBU) tests selected to measure core motor control of the gymnasts pre-intervention and post-intervention as they help evaluate core control in the three planes of motion. The units of measure are mmHg as the device is an inflatable pad that calculates the pressure the lumbo-pelvic-hip complex exerts over the instrument.
  The two tests were performed to both sides.
Core stability results on Core strenght and endurance | Up to 12 weeks
  Change from pre-test to post-test in core strenght and endurance results.
  Hip-bridge test is a core stability test used to evaluate the core strength and endurance of the subject. The unit of measure are (s).
  The test was performed to both sides.
Balance results from a force platform (Center of pressure area) | Up to 16 weeks
  Change of Center of pressure (COP) area from pre-test to post-test in balance results.
  A Romberg test variant, one leg stance test (OLST or SOLEC) was selected to evaluate the gymnasts balance as the gymnasts usually perform their balances over one leg. Eyes open and closed variants were also applied to be able to find more differences between groups. These tests were performed over a force platform, considered a gold standard tool for analysis of postural balance deficits, by means of valid parameters and stabilometry measures of confidence, such as center of pressure (COP) area. The unit of measure is (mm²).
Balance results from a force platform (Sway velocity) | Up to 16 weeks
  Change of sway velocity of the COP from pre-test to post-test in balance results.
  A Romberg test variant, one leg stance test (OLST or SOLEC) was selected to evaluate the gymnasts balance as the gymnasts usually perform their balances over one leg. Eyes open and closed variants were also applied to be able to find more differences between groups. These tests were performed over a force platform, considered a gold standard tool for analysis of postural balance deficits, by means of valid parameters and stabilometry measures of confidence, such as frequency and speed of displacement of the COP. The unit of measure is (mm/s).
Balance results from expert judging | Up to 16 weeks
  Change from pre-test to post-test in balance results.
  Three RG specific balances were selected to evaluate the execution and more specific balance technique of the gymnasts. Pase balance, side balance with help and arabesque balance were performed over the force platform and evaluated by RG international judges experts. The units of measure were points given from the judges.
Jump results from a force platform (height) | Up to 14 weeks
  Change of height from pre-test to post-test in jump results.
  Counter movement jump (CMJ) and single leg counter movement jump (SLCMJ) tests are selected to evaluate gymnasts' jump parameters. Gymnasts perform their leaps with the impulse of one or two legs, thus, it is important to evaluate jumps tests performed from one and both legs. The unit of measure is (m).
Jump results from a force platform (speed) | Up to 14 weeks
  Change speed from pre-test to post-test in jump results.
  Counter movement jump (CMJ) and single leg counter movement jump (SLCMJ) tests are selected to evaluate gymnasts' jump parameters. Gymnasts perform their leaps with the impulse of one or two legs, thus, it is important to evaluate jumps tests performed from one and both legs. The unit of measure is (m/s)
Jump results from a force platform (time of flight) | Up to 14 weeks
  Change of time of flight from pre-test to post-test in jump results.
  Counter movement jump (CMJ) and single leg counter movement jump (SLCMJ) tests are selected to evaluate gymnasts' jump parameters. Gymnasts perform their leaps with the impulse of one or two legs, thus, it is important to evaluate jumps tests performed from one and both legs. The unit of measure is (s).
Jump results from a force platform (power) | Up to 14 weeks
  Change of power from pre-test to post-test in jump results.
  Counter movement jump (CMJ) and single leg counter movement jump (SLCMJ) tests are selected to evaluate gymnasts' jump parameters. Gymnasts perform their leaps with the impulse of one or two legs, thus, it is important to evaluate jumps tests performed from one and both legs. The unit of measure is (W).
Jump results from a force platform (force) | Up to 14 weeks
  Change of force from pre-test to post-test in jump results.
  Counter movement jump (CMJ) and single leg counter movement jump (SLCMJ) tests are selected to evaluate gymnasts' jump parameters. Gymnasts perform their leaps with the impulse of one or two legs, thus, it is important to evaluate jumps tests performed from one and both legs. The unit of measure is (N).
Jump results from expert judging | Up to 14 weeks
  Change from pre-test to post-test in jump results.
  Three RG specific jump elements with different techniques were selected to be evaluated by RG international judges experts, these are the scissors, the stag and the split leap. The units of measure were points given from the judges.

SECONDARY OUTCOMES:
The Borg Rating of Perceived Exertion (RPE) scale | up to 8 weeks
  In order to regulate the intensity of the Core Stability Training the Borg Scale was used. The specific training load was calculated with the RPE session (Foster et al., 2001). The intensity of the training was aimed to be between 7-8 in the Borg Cr10 Scale. This scale value was selected as an outcome regarding the correct execution of the exercises and promoting training adaptations.
  Minimum and maximum values of the Borg Cr10 Scale, with the lowest values being the less intense workouts and the highest values being physical activity with very hard and maximum intensity
  Score and level of exertion:
  0- No exertion at all, 0.5- Very, very slight (just noticeable), 1- Very slight, 2- Slight ,3- Moderate, 4- Somewhat severe, 5- Severe, 6, 7, 8- Very severe, 9- Very, very severe (almost maximal), 10- Maximal
Peak height velocity (PHV) age | up to 16 weeks
  To ensure the results are not conditioned by group differences regarding maturity age, peak height velocity (PHV) of the gymnasts was calculated.
  Using the anthropometric measures in a multiple regression equation, the age of PHV was predicted. The outcome is measured in years and it represents the year where the gymnasts achieve the fastest upward growth in their stature.
Years from PHV age | up to 16 weeks
  To ensure the results are not conditioned by group differences regarding maturity age and to be able to place each gymnast in their maturing stage, years from peak height velocity (PHV) were calculated.
  Using the anthropometric measures in a multiple regression equation, the years from PHV were predicted. The equation calculates the time interval in years between the predicted age at PHV and the individual's current age; the values can be negative (the age of PHV not yet reached), positive (the age of PHV has passed) or zero (0) (the current age is the exact age of PHV).

CONTACTS AND LOCATIONS:
Locations (1):
- Blanquerna FPCEE, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panjabi MM. The stabilizing system of the spine. Part I. Function, dysfunction, adaptation, and enhancement. J Spinal Disord. 1992 Dec;5(4):383-9; discussion 397. doi: 10.1097/00002517-199212000-00001. PMID 1490034
- [Background] Kibler WB, Press J, Sciascia A. The role of core stability in athletic function. Sports Med. 2006;36(3):189-98. doi: 10.2165/00007256-200636030-00001. PMID 16526831
- [Background] Akuthota V, Nadler SF. Core strengthening. Arch Phys Med Rehabil. 2004 Mar;85(3 Suppl 1):S86-92. doi: 10.1053/j.apmr.2003.12.005. PMID 15034861
- [Background] McGill, S. (2010). Core training: Evidence translating to better performance and injury prevention. Strength & Conditioning Journal, 32(3), 33-46.
- [Background] Hibbs AE, Thompson KG, French D, Wrigley A, Spears I. Optimizing performance by improving core stability and core strength. Sports Med. 2008;38(12):995-1008. doi: 10.2165/00007256-200838120-00004. PMID 19026017
- [Background] Leetun DT, Ireland ML, Willson JD, Ballantyne BT, Davis IM. Core stability measures as risk factors for lower extremity injury in athletes. Med Sci Sports Exerc. 2004 Jun;36(6):926-34. doi: 10.1249/01.mss.0000128145.75199.c3. PMID 15179160
- [Background] Lederman E. The myth of core stability. J Bodyw Mov Ther. 2010 Jan;14(1):84-98. doi: 10.1016/j.jbmt.2009.08.001. PMID 20006294
- [Background] Azevedo DC, Lauria AC, Pereira AR, Andrade GT, Ferreira ML, Ferreira PH, Van Dillen L. Intraexaminer and interexaminer reliability of pressure biofeedback unit for assessing lumbopelvic stability during 6 lower limb movement tests. J Manipulative Physiol Ther. 2013 Jan;36(1):33-43. doi: 10.1016/j.jmpt.2012.12.008. PMID 23380212
- [Background] Mirwald RL, Baxter-Jones AD, Bailey DA, Beunen GP. An assessment of maturity from anthropometric measurements. Med Sci Sports Exerc. 2002 Apr;34(4):689-94. doi: 10.1097/00005768-200204000-00020. PMID 11932580
- [Background] Foster C, Florhaug JA, Franklin J, Gottschall L, Hrovatin LA, Parker S, Doleshal P, Dodge C. A new approach to monitoring exercise training. J Strength Cond Res. 2001 Feb;15(1):109-15. PMID 11708692
- [Background] Briggs RC, Gossman MR, Birch R, Drews JE, Shaddeau SA. Balance performance among noninstitutionalized elderly women. Phys Ther. 1989 Sep;69(9):748-56. doi: 10.1093/ptj/69.9.748. PMID 2772037
- [Background] da Silva RA, Bilodeau M, Parreira RB, Teixeira DC, Amorim CF. Age-related differences in time-limit performance and force platform-based balance measures during one-leg stance. J Electromyogr Kinesiol. 2013 Jun;23(3):634-9. doi: 10.1016/j.jelekin.2013.01.008. Epub 2013 Feb 10. PMID 23403137
- [Background] di Cagno A, Baldari C, Battaglia C, Guidetti L, Piazza M. Anthropometric characteristics evolution in elite rhythmic gymnasts. Ital J Anat Embryol. 2008 Jan-Mar;113(1):29-35. PMID 18491452
- [Background] Georgopoulos NA, Markou KB, Theodoropoulou A, Vagenakis GA, Mylonas P, Vagenakis AG. Growth, pubertal development, skeletal maturation and bone mass acquisition in athletes. Hormones (Athens). 2004 Oct-Dec;3(4):233-43. doi: 10.14310/horm.2002.11132. PMID 16982598
- [Background] Markovic G, Dizdar D, Jukic I, Cardinale M. Reliability and factorial validity of squat and countermovement jump tests. J Strength Cond Res. 2004 Aug;18(3):551-5. doi: 10.1519/1533-4287(2004)182.0.CO;2. PMID 15320660
- [Background] Miletic D, Katic R, Males B. Some anthropologic factors of performance in rhythmic gymnastics novices. Coll Antropol. 2004 Dec;28(2):727-37. PMID 15666605
- [Background] Donti O, Bogdanis GC, Kritikou M, Donti A, Theodorakou K. The relative contribution of physical fitness to the technical execution score in youth rhythmic gymnastics. J Hum Kinet. 2016 Jul 2;51:143-152. doi: 10.1515/hukin-2015-0183. eCollection 2016 Jun 1. PMID 28149377
- [Background] Douda HT, Toubekis AG, Avloniti AA, Tokmakidis SP. Physiological and anthropometric determinants of rhythmic gymnastics performance. Int J Sports Physiol Perform. 2008 Mar;3(1):41-54. doi: 10.1123/ijspp.3.1.41. PMID 19193953
- [Background] Baxter-Jones AD. Growth and development of young athletes. Should competition levels be age related? Sports Med. 1995 Aug;20(2):59-64. doi: 10.2165/00007256-199520020-00001. No abstract available. PMID 7481282
- [Background] Malina RM, Baxter-Jones AD, Armstrong N, Beunen GP, Caine D, Daly RM, Lewis RD, Rogol AD, Russell K. Role of intensive training in the growth and maturation of artistic gymnasts. Sports Med. 2013 Sep;43(9):783-802. doi: 10.1007/s40279-013-0058-5. PMID 23743792
- [Background] Asseman FB, Caron O, Cremieux J. Are there specific conditions for which expertise in gymnastics could have an effect on postural control and performance? Gait Posture. 2008 Jan;27(1):76-81. doi: 10.1016/j.gaitpost.2007.01.004. Epub 2007 Mar 6. PMID 17337190
- [Background] Calavalle AR, Sisti D, Rocchi MB, Panebianco R, Del Sal M, Stocchi V. Postural trials: expertise in rhythmic gymnastics increases control in lateral directions. Eur J Appl Physiol. 2008 Nov;104(4):643-9. doi: 10.1007/s00421-008-0815-6. Epub 2008 Jul 10. PMID 18618136
- [Background] Watson T, Graning J, McPherson S, Carter E, Edwards J, Melcher I, Burgess T. DANCE, BALANCE AND CORE MUSCLE PERFORMANCE MEASURES ARE IMPROVED FOLLOWING A 9-WEEK CORE STABILIZATION TRAINING PROGRAM AMONG COMPETITIVE COLLEGIATE Dancers. Int J Sports Phys Ther. 2017 Feb;12(1):25-41. PMID 28217414
- [Background] Liebenson C, Karpowicz AM, Brown SH, Howarth SJ, McGill SM. The active straight leg raise test and lumbar spine stability. PM R. 2009 Jun;1(6):530-5. doi: 10.1016/j.pmrj.2009.03.007. PMID 19627942

DOCUMENTS (1):
  • Informed Consent Form (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT04663633/ICF_000.pdf